CLINICAL TRIAL: NCT05702424
Title: An Open-Label, Multicenter, Phase 1 Study of IGM-7354 in Adult Participants With Relapsed and/or Refractory Cancer
Brief Title: Evaluation of IGM-7354 in Adults With Relapsed and/or Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IGM-7354-001
Record Dates: First submitted 2023-01-13; First posted 2023-01-27 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumor
Keywords: Relapsed and/or Refractory; Metastatic Cancer; Advanced Tumors; Incurable
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IGM-7354 Single-Agent Dose Escalation (Experimental): IGM-7354 will be administered intravenously as a single agent.
  Interventions: Drug: IGM-7354
- IGM-7354 Single-Agent Dose Expansion Serial Biopsy (Experimental): IGM-7354 will be administered intravenously as a single agent and patients will undergo pre-treatment and on-treatment biopsies.
  Interventions: Drug: IGM-7354

INTERVENTIONS:
Drug: IGM-7354 — IGM-7354 is a PD-L1-targeted cytokine that is designed to regulate T and natural killer cell activation, proliferation and promote their anti-tumor effects

SUMMARY:
This study is a first-in-human (FIH), Phase 1, multicenter, open-label study to evaluate the safety, tolerability, and PK of IGM-7354 in participants with relapsed and/or refractory tumors. The study design consists of a dose-escalation stage and dose-expansion stage. Study participation will consist of a 28-day screening period, a treatment period, and a safety follow-up period 90-days after the last dose.

DETAILED DESCRIPTION:
Patients will be enrolled in two stages: a dose-escalation stage and an expansion stage. The escalation stage will investigate single agent IGM-7354 safety and tolerability in patients with relapsed and/or refractory solid tumors. The dose expansion serial biopsy cohort will assess the intra-tumoral PD changes related to the activity of IGM-7354.

IGM-7354 will be administered intravenously (IV).

ELIGIBILITY:
Key Inclusion Criteria:

* Age > 18 years at time of signing ICF
* ECOG Performance Status of 0 or 1
* Histologic or cytologic documentation of incurable, locally advanced or metastatic solid tumors for which standard therapies are not available, are no longer effective, are not tolerated, or have been declined by the participant
* Participants with either measurable or evaluable disease
* Adequate organ function
* At least 2 weeks prior to Day 1 or 5 half-lives, whichever is shorter, must have elapsed from the use of anti-tumor therapy, including chemotherapy, biologic, experimental, or hormonal therapy
* Participants must be willing to have pre-treatment and on-treatment tumor biopsies for biomarker evaluation

Key Exclusion Criteria:

* Inability to comply with study and follow-up procedures
* Prior IL-15, IL-2, synthetic IL-2, or IL-2v based therapy
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Palliative radiation to bone metastases within 2 weeks prior to Day 1
* Major surgical procedure within 4 weeks prior to Day 1
* Untreated or active central nervous system (CNS) metastases. Patients with a history of treated CNS metastases are eligible.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* Diagnosis of immunodeficiency
* Current Grade >1 toxicity from prior therapy. Participants with current Grade 2 chronic toxicities that are well-controlled by medications may be enrolled after discussion with medical monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of IGM-7354 in participants with cancer including estimation of the MTD or MAD | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 12 months (each cycle is 28 days)
  Incidence of treatment-emergent AEs, SAEs, and DLT per NCI CTCAE v5.0

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of IGM-7354 | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 12 months (each cycle is 28 days)
  Area Under the Curve (AUC) of IGM-7354 as a single agent
Clearance (CL) of IGM-7354 | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 12 months (each cycle is 28 days)
  Clearance (CL) of IGM-7354 as a single agent
Volume of distribution (V) of IGM-7354 | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 12 months (each cycle is 28 days)
  Volume of distribution (V) of IGM-7354 as a single agent
Maximum Plasma Concentration (Cmax) of IGM-7354 | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 12 months (each cycle is 28 days)
  Maximum Plasma Concentration (Cmax) of IGM-7354 as a single agent
Objective Response Rate (ORR) | Study duration of approximately 29 months
  The ORR is defined as the percentage of participants who achieve a confirmed complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by investigators
Duration of Response (DoR) | Study duration of approximately 29 months
  For participants who demonstrate confirmed CR or PR, duration of response is defined as the time from the first documented CR or PR to the first documented disease progression or death, whichever occurs first.
Progression-Free Survival (PFS) | Study duration of approximately 29 months
  PFS is defined as the time from first dose to the first documented disease progression per RECIST 1.1 by investigator or death, whichever occurs first.
Anti-drug antibodies (ADAs) of IGM-7354 | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 12 months (each cycle is 28 days)
  Immunogenicity of IGM-7354

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — IGM Biosciences
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Oklahoma University, Norman, Oklahoma
  - START South Texas Accelerated Research Therapeutics, San Antonio, Texas